CLINICAL TRIAL: NCT02895074
Title: Subfoveal Choroidal Thickness After Femtosecond Laser-assisted Cataract Surgery for Age-related Cataracts
Brief Title: Subfoveal Choroidal Thickness After Surgery for Age-related Cataracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2016-China7
Record Dates: First submitted 2016-08-29; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Cataract
Keywords: femtosecond laser-assisted cataract surgery (FLACS); subfoveal choroidal thickness (SFCT); conventional phacoemulsification surgery (CPS)
MeSH Terms: conditions — Cataract | interventions — Tropicamide; proxymetacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- femtosecond laser-assisted cataract surgery group (Experimental)
  Interventions: Procedure: Femtosecond laser-assisted cataract surgery; Drug: Tropicamide; Drug: Proparacaine hydrochloride
- conventional phacoemulsification surgery group (Experimental)
  Interventions: Procedure: Conventional phacoemulsification cataract surgery; Drug: Tropicamide; Drug: Proparacaine hydrochloride

INTERVENTIONS:
Procedure: Femtosecond laser-assisted cataract surgery — A femtosecond laser (Alcon-Lensx, Alcon-Lensx, Inc.) was used in this study. After pupil dilation and topical anesthesia, the laser was docked to the eye using a curved contact lens to applanate the cornea. With the integrated OCT imaging system, the locations of the cornea and the anterior and posterior surfaces of the crystalline lens were determined. A 5.0-mm-diameter capsulotomy was created by scanning a cylindrical pattern and followed by lens fragmentation. The laser was disconnected, and the remainder of the surgery was performed as phacoemulsification (Infiniti® Vision System; Alcon, USA). Folded intraocular lenses (IOLs) were implanted in the capsular bags.
  Arms: femtosecond laser-assisted cataract surgery group
Procedure: Conventional phacoemulsification cataract surgery — Phacoemulsification was performed through a temporal 3.2-mm clear corneal incision with the same machine and followed by IOLs implantation.
  Arms: conventional phacoemulsification surgery group
Drug: Tropicamide — After pupil dilation, 1 drop of tropicamide (0.5%) was applied every 15 minutes for 3 applications
Drug: Proparacaine hydrochloride — topical anesthesia with proparacaine hydrochloride (0.5%) was applied.

SUMMARY:
To compare the effects of femtosecond laser-assisted cataract surgery (FLACS) and conventional phacoemulsification surgery (CPS) on subfoveal choroidal thickness (SFCT) in age-related cataracts.

DETAILED DESCRIPTION:
It is not clear whether femtosecond laser-assisted cataract surgery (FLACS) alters retinal and choroidal thickness. The goal of the present study was to determine the changes of retinal and choroidal thicknesses in patients who have undergone FLACS compared to patients who have undergone conventional phacoemulsification surgery (CPS).

ELIGIBILITY:
Inclusion Criteria:

* The cataract stages of the patients were between N2 and N4 according to the LOCS III.

Exclusion Criteria:

* eyes with histories of ocular surgery, trauma, and ocular diseases, including diabetic retinopathy, age-related macular degeneration (AMD), high myopia, psudoexfoliation, uveitis, retinal vein occlusion, and other inflammatory and vascular retinal disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The change of subfoveal choroidal thickness | baseline, at 1 day after surgery, 7 days after surgery, 1 month after surgery, and 3 months after surgery
  The subfoveal choroidal thickness were measured at baseline and at 1 day, 7 days , 1 month , and 3 months postoperatively by spectral-domain optical coherence tomography.

SECONDARY OUTCOMES:
The change of subfoveal retinal thickness | baseline, at 1 day after surgery, 7 days after surgery, 1 month after surgery, and 3 months after surgery
  The subfoveal retinal thickness were measured at baseline and at 1 day, 7 days , 1 month , and 3 months postoperatively by spectral-domain optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen X, Xiao W, Ye S, Chen W, Liu Y. Efficacy and safety of femtosecond laser-assisted cataract surgery versus conventional phacoemulsification for cataract: a meta-analysis of randomized controlled trials. Sci Rep. 2015 Aug 13;5:13123. doi: 10.1038/srep13123. PMID 26269445
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/
- See also: Homepage of Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH) — http://www.cnccclub.com/